CLINICAL TRIAL: NCT02608931
Title: The Safety , Tolerability and Efficacy of Dronabinol, a Synthetic Endocannabinoid Receptor Agonist, for the Treatment of Nausea and Vomiting in Patients With Familial Dysautonomia
Brief Title: The Safety, Tolerability and Efficacy of Dronabinol, for the Treatment of Nausea and Vomiting in Familial Dysautonomia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to begin study with drug provider
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14-01577
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Nausea; Vomiting; Familial Dysautonomia
Keywords: delta-9-tetrahydrocannabinol (THC)
MeSH Terms: conditions — Nausea; Vomiting; Dysautonomia, Familial | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dranabinol Capsules (Experimental): The initial dose will be 2.5 mg BID (5 mg/day), and the maximum dose will be 10 mg TID (30 mg/day).
  Interventions: Drug: Dronabinol
- Placebo Capsules (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dronabinol
  Other Names: Marinol
  Arms: Dranabinol Capsules
Other: Placebo — placebo
  Arms: Placebo Capsules

SUMMARY:
This is a pilot clinical trial of dronabinol to treat disabling attacks of nausea and vomiting in patients with familial dysautonomia (FD, also known as Riley Day syndrome or hereditary sensory and autonomic neuropathy type III). FD is a rare autosomal recessive disease in which the growth and development of selective nerves is impaired. Patients with FD suffer recurrent uncontrollable nausea and vomiting crises accompanied by skin flushing, tachycardia and arterial hypertension. Current treatments of nausea are ineffective or have intolerable side sides. Our long-term goal is to treat nausea effectively and without side effects, a therapeutic intervention that would markedly improve the quality of life of patients with FD.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the safety, tolerability and efficacy of dronabinol for the treatment of nausea in patients with FD. The pilot trial will recruit 25 patients with FD who complain of severe nausea that affects their quality of life. The trial will be divided into two consecutive, but independent parts. Part 1, will address the safety and tolerability of dronabinol in patients with FD using an open-label dose titration phase followed by 4-weeks of wash-out period. Part 2 will address the efficacy of dronabinol for the treatment of nausea in patients with FD using a randomized, placebo controlled, double blind, 12-week cross over design.

The first specific aim of this proposal is to assess the safety and tolerability of dronabinol in patients with FD. The second specific aim of this proposal is to determine whether stimulation of endocannabinoid receptors with dronabinol will improve recurrent nausea in patients with FD. Secondary aims are to determine whether stimulation of endocannabinoid receptors with dronabinol will increase weight, and decrease anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-60.
2. Confirmed diagnosis of familial dysautonomia by genetic testing.
3. Symptoms of severe nausea.
4. Able to swallow the capsules.
5. Written informed consent or ascent to participate in the pilot trial and understanding that they can withdraw consent or accent at anytime without affecting their future care.
6. Ability to comply with the requirements of the study procedures, including taking blood pressure measurements at home

Exclusion Criteria:

1. Patients with a history of hypersensitivity to any cannabinoid or sesame oil.
2. Cannabinoid use in the previous 4 weeks (a urinary cannabinoid test will be performed before study entry).
3. Patients with a history of substance abuse, including alcohol abuse or dependence, or marijuana.
4. Seizure disorder with at least one epileptic seizure in the last 3 years or abnormal epileptic discharge in electroencephalography
5. Patients with history of bipolar disorder, severe depression or schizophrenia.
6. Patients that require driving, operating machinery, or engaging in hazardous activities.
7. Patients taking medications thought, in the investigator's opinion, to be unsafe when used with dronabinol.
8. Patients with atrial fibrillation, angina or an electrocardiogram documenting a significant abnormality that may jeopardize the patient's health.
9. Patients with significant pulmonary, liver, renal (creatinine > 2.0 mg/ml), or cardiac illness that may, in the investigators opinion jeopardize their health by participating in this pilot trial.
10. Patients with severe cognitive impairment or pervasive developmental disorders, or patients who are unable to clearly identify and rate their symptoms of nausea.
11. Women who are pregnant or lactating.
12. Patients who have a significant abnormality on clinical examination that may, in the investigator's opinion, jeopardize their health by participating in this pilot trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Number of adverse effects | 8 weeks
  number of AEs during 4 weeks active drug phase vs. 4 weeks placebo phase
Change in nausea scores | 8 weeks
  nausea scores during 4 weeks active drug phase vs. 4 weeks placebo phase

SECONDARY OUTCOMES:
Change in weight. | 8 weeks
  change in weight (kgs) during 4 weeks active drug phase vs. 4 weeks placebo phase
Change in anxiety scores | 8 Weeks
  change in anxiety scale scores during 4 weeks active drug phase vs. 4 weeks placebo

CONTACTS AND LOCATIONS:
Overall Officials: Horacio C Kaufmann, MD, Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- NYU Medical Center, New York, New York, United States